CLINICAL TRIAL: NCT02705131
Title: Balance Chiropractic Therapy for Cervical Spondylotic Radiculopathy: a Randomized Parallel-controlled Trial
Brief Title: Balance Chiropractic Therapy for Cervical Spondylotic Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Feng Yang (Other)
Responsible Party: Sponsor-Investigator, Feng Yang, Principal Investigator, Shaanxi University of Chinese Medicine
Organization: Shaanxi University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SXUCM-018
Record Dates: First submitted 2016-02-28; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical radiculopathy; Balance chiropractic therapy
MeSH Terms: conditions — Radiculopathy | interventions — Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Chiropractic Therapy(BCT) (Experimental): patients are in the sitting position and receive the Balance Chiropractic Therapy(BCT) .1)Balancing tendon-regulation;2) Balancing osteopathy;3) Balance collaterals-dredging.The patients will received BCT 1 time every other day, 20min each time. a total of 10 times in 20 days.
  Interventions: Device: Balance Chiropractic Therapy
- Traction Therapy(TT) (Active Comparator): patients will receive the Traction Therapy(TT):The patient is sitting and wearing a cloth bag occipital jaw traction comfortable,with head bending forward about 10-15 degrees in comfort.The weight for traction of cervical spondylosis is started at 3 kg, and gradually increased to the maximum weight not more than 6kg according to the standard of 0.5kg each time. The treatment is performed 30 minutes a time per day, 10 times as a course,a total of 2 courses.
  Interventions: Device: Traction Therapy

INTERVENTIONS:
Device: Balance Chiropractic Therapy — patients are in the sitting position and receive the following treatments.1)Balancing tendon-regulation;2) Balancing osteopathy;3) Balance collaterals-dredging.
  Arms: Balance Chiropractic Therapy(BCT)
Device: Traction Therapy — patients will received the traction therapy.The patient is sitting and wearing a cloth bag occipital jaw traction comfortable,with head bending forward about 10-15 degrees in comfort.The weight for traction of cervical spondylosis is started at 3 kg, and gradually increased to the maximum weight not more than 6kg according to the standard of 0.5kg each time. The treatment is performed 30 minutes a time per day, 10 times as a course,a total of 2 courses.
  Arms: Traction Therapy(TT)

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect and safety of the Balance Chiropractic Therapy(BCT) on Cervical Spondylotic Radiculopathy and to investigate the mechanism of which this efficacy is achieved.

DETAILED DESCRIPTION:
The investigators propose a multi center randomized, parallel-controlled trial to evaluate the efficacy and safety of the balance chiropractic therapy for CSR. Participants aged 18 to 65, who are in conformity with the diagnostic criteria of CSR and the pain score regarding visual analog scales is more than 4 points and less than 8 points, will be included and randomly allocated into two groups: test group and control group. Participants in the test group will be treated with the balance chiropractic therapy, while the control group will receive the traction therapy. The primary outcome is pain severity (measured with a visual analogue scale (VAS)). Secondary outcomes will include cervical curvature (measured by Borden index), a composite of functional status(measured by Neck Disability Index ,NDI), individual patients health status(evaluated by SF-36 health survey ), and adverse events as reported in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are in conformity with the diagnostic criteria of CSR;
* Aged between18 and 65 years old;
* The pain score regarding visual analog scales is more than 4 points and less than 8 points;
* sign the informed consent.

Exclusion Criteria:

* Subjects will be excluded if they have disorders such as vague diagnosis of acute spinal cord injury or acute spinal cord inflammation,or cervical vertigo symptom and checking for abnormal changes on transcranial doppler(TCD).
* Subjects will also be excluded if they have combined liver, kidney, hematopoietic system, endocrine system, cardiovascular system, nervous system and other severe primary disease,or fractures,osteoarticular tuberculosis, osteomyelitis, bone tumor, severe osteoporosis,or mental disabilities,
* A weak body can not withstand the stimulation of the balance chiropractic therapy .
* Individuals who have acute infectious disease, stomach or duodenal ulcer with acute perforation,or treated areas with severe skin damage or skin diseases.
* Subjects that have received surgical treatment or neck injury, or radiofrequency of cervical intervertebral disc, or minimally invasive, or ozone, or acupuncture and moxibustion, or other manipulations or block therapy within two weeks
* Lactating or pregnant patients.
* Subjects who are participating in other clinical trials related to cervical spondylosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Pain Scores as measured by the Visual Analog Scale | Three months

SECONDARY OUTCOMES:
cervical curvature as measured by Borden method | three months
composite of functional status as measured by Neck Disability Index | three months
Health Related Quality of Life as measured by SF-36 | three months

CONTACTS AND LOCATIONS:
Overall Officials: Li Liu, Dr., Study Chair — Shaanxi university of TCM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campa-Moran I, Rey-Gudin E, Fernandez-Carnero J, Paris-Alemany A, Gil-Martinez A, Lerma Lara S, Prieto-Baquero A, Alonso-Perez JL, La Touche R. Comparison of Dry Needling versus Orthopedic Manual Therapy in Patients with Myofascial Chronic Neck Pain: A Single-Blind, Randomized Pilot Study. Pain Res Treat. 2015;2015:327307. doi: 10.1155/2015/327307. Epub 2015 Nov 10. PMID 26640708
- [Result] Tanaka Y, Kokubun S, Sato T, Ozawa H. Cervical roots as origin of pain in the neck or scapular regions. Spine (Phila Pa 1976). 2006 Aug 1;31(17):E568-73. doi: 10.1097/01.brs.0000229261.02816.48. PMID 16924193
- [Result] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Result] Carlin JB, Doyle LW. Sample size. J Paediatr Child Health. 2002 Jun;38(3):300-4. doi: 10.1046/j.1440-1754.2002.00855.x. No abstract available. PMID 12047701
- [Result] Binder AI. Cervical spondylosis and neck pain. BMJ. 2007 Mar 10;334(7592):527-31. doi: 10.1136/bmj.39127.608299.80. No abstract available. PMID 17347239
- [Derived] Li W, Chang Y, Feng Q, Cheng Y, Yin J, Sun Y, Yang F. Balance chiropractic therapy for cervical spondylotic radiculopathy: A randomized controlled trial. Contemp Clin Trials Commun. 2024 Jul 14;41:101323. doi: 10.1016/j.conctc.2024.101323. eCollection 2024 Oct. PMID 39188412
- [Derived] Yang F, Li WX, Liu Z, Liu L. Balance chiropractic therapy for cervical spondylotic radiculopathy: study protocol for a randomized controlled trial. Trials. 2016 Oct 22;17(1):513. doi: 10.1186/s13063-016-1644-2. PMID 27770801